CLINICAL TRIAL: NCT06282263
Title: The Effect of the Awareness Development Program on Suicide Prevention for Oncology Nurses on the Levels of Suicide Knowledge, Stigma and Perception of Efficacy
Brief Title: The Effect of the Awareness Development Program on Suicide Prevention for Oncology Nurses
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sevda Ozturk (Other)
Responsible Party: Sponsor-Investigator, Sevda Ozturk, Research Assistant Sevda Öztürk, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1292
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Suicide Prevention; Nurses
Keywords: suicide prevention; oncology
MeSH Terms: conditions — Suicide Prevention; Neoplasms

STUDY DESIGN:
Intervention Model Description: This study was a pre-test, post-test, follow-up design and control group intervention study conducted to examine the effect of "Awareness Development Programme on Suicide Prevention for Oncology Nurses" on oncology nurses' knowledge, stigma and perception of efficacy regarding suicide risk management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): "Awareness Development Program on Suicide Prevention for Oncology Nurses" was applied to the nurses in the experimental group.
  Interventions: Other: "Awareness Development Program on Suicide Prevention for Oncology Nurses"
- Control Group (No Intervention): No programme was applied to the control group.

INTERVENTIONS:
Other: "Awareness Development Program on Suicide Prevention for Oncology Nurses" — While developing the "Awareness Development Programme on Suicide Prevention for Oncology Nurses" applied to the nurses in the experimental group, literature information on suicide risk management and suicide prevention in oncology was included in the study content by the researchers. "Awareness Development Programme on Suicide Prevention for Oncology Nurses" includes 3 sessions and the titles of the programme are as follows:
  Session 1: Introduction to Understanding Suicide "Awareness and Development" Session 2: Assessing Suicide Risk Session 3: Management of Suicide Risk "Communication and Referral" The programme was submitted to the opinions of 5 experts before starting the study and the programme was finalised after the feedbacks.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to investigate the effect of the Awareness Development Programme on Suicide Prevention for Oncology Nurses on the levels of knowledge, stigma and perception of efficacy towards suicide in oncology nurses. The main questions it aims to answer are:

1. At the end of the Awareness Development Programme on Suicide Prevention for Oncology Nurses applied to nurses working in the field of oncology and at the end of the 3-month follow-up, is there a difference between the knowledge levels of nurses about suicide according to the pre-programme and control group?
2. At the end of the Awareness Development Programme on Suicide Prevention for Oncology Nurses applied to nurses working in the field of oncology and at the end of the 3-month follow-up, is there a difference between the perception of efficacy levels of nurses regarding suicide according to the pre-programme and control group.
3. At the end of the Awareness Development Programme on Suicide Prevention for Oncology Nurses applied to nurses working in the field of oncology and at the end of the 3-month follow-up, is there a difference between the stigma levels of nurses towards suicide according to the pre-programme and control group.
4. Is there a significant relationship between the levels of knowledge about suicide, perception of efficacy regarding suicide, and stigma towards suicide in the pre-test and post-test measurements of the Awareness Development Programme on Suicide Prevention for Oncology Nurses applied to nurses working in the field of oncology.
5. Is there a significant relationship between the levels of knowledge about suicide, perception of efficacy regarding suicide, and stigma towards suicide in the pre-test-follow-up test measurements of the Awareness Development Programme on Suicide Prevention for Oncology Nurses applied to nurses working in the field of oncology.

Participants will participate the Awareness Development Programme on Suicide Prevention for Oncology Nurses. Oncology Nurses are expected to complete the pre-test, post-test and follow-up tests.

Researchers will compare control group to see if effect of "the Awareness Development Programme on Suicide Prevention"

DETAILED DESCRIPTION:
This research is an intervention study with a pre-test, post-test, follow-up design and control group, which was conducted to examine the effect of the "Awareness Development Program on Suicide Prevention for Oncology Nurses" on oncology nurses' knowledge, stigma and effectiveness perception levels regarding managing suicide risk.

ELIGIBILITY:
Inclusion Criteria:

* To be willing to participate in the study,
* Being a nurse working in oncology inpatient clinics (medical oncology, medical oncology, gastroenterology oncology, nephrology oncology, urooncology, gynaecological oncology, haematological oncology inpatient clinics), Bone Marrow Transplantation (BMT) unit, outpatient chemotherapy unit and oncology outpatient clinic,
* To know how to use a smart mobile phone or computer.

Exclusion Criteria:

* To have training other than undergraduate education for suicide prevention,
* To care for paediatric oncology patients,
* To have worked in a psychiatric clinic or to have postgraduate education in the field of psychiatric nursing.
* Failure to attend two out of three sessions during the training programme,
* Failure to demonstrate the motor skills to participate in online training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
the Literacy of Suicide Scale | Pretests were applied before the sessions. Intervention sessions of three sessions were implemented 5-8 days apart. Post-tests were administered as soon as the third session was completed. Follow-up tests were conducted 90 days after the post-tests.
  A minimum score of 0 and a maximum total score of 27 can be obtained from the scale. The scale does not have any cut-off point. The higher the score obtained from the scale, the higher the level of knowledge about suicide.
Efficacy Perception Scale For Suicide Risk Management | Pretests were applied before the sessions. Intervention sessions of three sessions were implemented 5-8 days apart. Post-tests were administered as soon as the third session was completed. Follow-up tests were conducted 90 days after the post-tests.
  This scale consists of 26 items. The lowest score that can be obtained from this scale is 26 and the highest score is 130, and the scale has no cut-off point. An increase in the score obtained from the scale indicates that nurses' self-perception is becoming more positive in relation to their knowledge and skills in the recognition and management of suicide risk.
The Stigma of Suicide Scale | Pretests were applied before the sessions. Intervention sessions of three sessions were implemented 5-8 days apart. Post-tests were administered as soon as the third session was completed. Follow-up tests were conducted 90 days after the post-tests.
  There are 55 items in total in the scale. The scale has three subscales: "stigma", "isolation/depression" and "glorification/normalization". Total score is not calculated in the scale. High scores from the "stigma" sub-dimension of the scale indicate high stigma towards suicide. High scores from the "isolation/depression" sub-dimension of the scale indicate that suicide is more associated with depression and isolation, while high scores from the "normalization" sub-dimension indicate that individuals normalize suicide rather than stigmatizing people who commit suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Hiçdurmaz, Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No